CLINICAL TRIAL: NCT01733095
Title: Ambrisentan for Treatment of Portopulmonary Hypertension (PoPH): a Pilot Study
Brief Title: Ambrisentan for Treatment of Portopulmonary Hypertension
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PoPH-GRZ ambrisentan
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Portopulmonary Hypertension
MeSH Terms: interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ambrisentan (Experimental): In all patients with clinically significant PoPH, ambrisentan will be administered orally using a low ascending dose regime (see below). Duration of treatment will be 12 months.
  Interventions: Drug: ambrisentan

INTERVENTIONS:
Drug: ambrisentan — Ambrisentan (Volibris 5 mg film-coated tablets, Glaxo Smith-Kline) will be started at 5 mg every other day and increased to 5 mg daily after 4 weeks if tolerated well.
  Other Names: Volibris

SUMMARY:
Portopulmonary hypertension denotes pulmonary hypertension complicating portal hypertension and is present in approximately 5% of cirrhotic patients. Treatment options include prostanoids, sildenafil, and the endothelin-receptor antagonists, bosentan and ambrisentan.

This study investigates the safety and efficacy of ambrisentan in portopulmonary hypertension.

DETAILED DESCRIPTION:
Patients with clinically significant PoPH (resting mean pulmonary arterial pressure >25 mm Hg, pulmonary vascular resistance >400 dynes*s*cm-5) will be offered treatment with ambrisentan. Patients will be followed clinically and hemodynamically up to 12 months after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with portal hypertension, age >18 years
* Cirrhosis of any etiology; Child-Pugh class A and B
* Noncirrhotic portal hypertension (e.g. chronic portal vein thrombosis)
* Informed consent

Exclusion Criteria:

* Presence of other causes for pulmonary arterial hypertension
* History of pulmonary embolism or myocardial infarction within 6 months before study start
* Child-Pugh class C
* Presence of hepatocellular carcinoma
* Liver transplantation
* HIV infection
* Severe obstructive or restrictive pulmonary disease (predicted FEV1 or VC <65%, respectively)
* Severe dilated cardiomyopathy (EF <50%)
* Latent left-heart insufficiency
* Pregnancy and lactation
* Esophageal variceal hemorrhage within the last 6 months
* Refractory ascites
* Hepatorenal syndrome
* Persistent hepatic encephalopathy > grade 1
* Bilirubin >3.0 mg/dl
* AST and/or ALT >3x ULN
* Creatinine >2.0 mg/dl
* Known hypersensitivity to ambrisentan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
pulmonary vascular resistance | week 24

SECONDARY OUTCOMES:
mean arterial pulmonary pressure | week 24
hepatic venous pressure gradient | week 24
exercise capacity | week 24, 48
quality of life | week 24, 48

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf E. Stauber, MD, Principal Investigator — Gastroenterology & Hepatology; Horst Olschewski, MD, Study Director — Pulmonology
Locations (1):
- Medical University of Graz, Graz, Austria